CLINICAL TRIAL: NCT02181725
Title: Effectiveness and Cost-effectiveness of a Multimodal Rehabilitation Programme (MRP) for Adolescents With Chronic Musculoskeletal Pain (12-21 Years) Compared to Care as Usual (CAU); a Randomized Clinical Trial (2B Active)
Brief Title: 2B Active: Outpatient Rehabilitation for Adolescents With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Fonds NutsOhra (Other); Stichting Vooruit (Unknown); Adelante, Centre of Expertise in Rehabilitation and Audiology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL47323.068.13/METC13-3-062; 1202-068 (Other Grant/Funding Number: Fonds NutsOhra)
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Adolescent; Graded Exposure
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal Rehabilitation Program (Experimental): Multimodal Rehabilitation Program, consisting of a Graded Exposure Module (GE), a Combination Module (HMGE) and a Parent Module (PM)
  Interventions: Behavioral: Multimodal Rehabilitation Program
- Care as Usual (Active Comparator): Care as usual is the care currently provided to adolescents with musculoskeletal chronic pain and is based on the principles of Graded Activity.
  Interventions: Behavioral: Care as Usual

INTERVENTIONS:
Behavioral: Multimodal Rehabilitation Program — The Multimodal Rehabilitation Program is a Graded exposure based treatment. It consists of a Graded Exposure Module (GE), a Combination Module (HMGE) and a Parent Module (PM).
  Other Names: MRP
  Arms: Multimodal Rehabilitation Program
Behavioral: Care as Usual — Care as usual is the care currently provided to adolescents with musculoskeletal chronic pain and is based on the principles of Graded Activity.
  Other Names: CAU
  Arms: Care as Usual

SUMMARY:
The purpose of this study is to evaluate whether a multimodal rehabilitation program effectively reduces functional disability in adolescents with chronic musculoskeletal pain, compared to care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-21 years at the start of the study
* Complaints of chronic non-specific musculoskeletal pain of a duration > 3 months
* Considerable activity limitations
* Fear of movement
* Indication for outpatient multidisciplinary rehabilitation treatment
* Adequate Dutch literacy to complete the assessments (which mainly comprise questionnaires)

Exclusion Criteria:

* Any suspicion of a medical (orthopaedic, rheumatic or neurological) disease, that can explain the current pain complaints
* Any suspicion of an (underlying) psychiatric disease, for which psychiatric treatment is better suited, according to the expert opinion of the consultant in rehabilitation medicine.
* Pregnancy

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change in Functional Disability | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported functional disability

SECONDARY OUTCOMES:
Change in Quality of life | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported pain-specific quality of life
Change in Fear of Pain | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported fear of pain
Change in Fear of Pain | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Parent proxy report measure
Change in Pain Catastrophizing | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported pain catastrophizing
Change in Pain Catastrophizing | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Parental catastrophizing about their child's pain
Change in Depressive symptoms | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported depressive symptoms
Change in Perceived Harmfulness | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported perceived harmfulness of daily activities
Change in Pain Intensity | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-reported pain intensity
Change in Functional Disability | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Parent-perceived functional disability of their child
Change in parental responses to childrens pain | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
Treatment expectations | Baseline
  Adolescent self-report
Treatment expectations | Baseline
  Parent self-report
Treatment satisfaction/ patient centeredness | 16 weeks
Treatment satisfaction/ family centeredness | 16 weeks
Change in General Health Related Quality of Life | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
Cost-diary per month | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Adolescent self-report of total health care utilization and other costs
Cost-diary per month | Baseline, 8 weeks, 16 weeks, 10 months, 12 months
  Parent self-reported adolescent related costs

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Goossens, PhD, Principal Investigator — Maastricht University, FHML, Department of Rehabilitation Medicine
Locations (4):
- Netherlands (4):
  - Maastricht University Medical Center, Maastricht, Limburg
  - Laurentius Ziekenhuis Roermond, Roermond, Limburg
  - Revant Revalidatiecentrum Breda, Breda, North Brabant
  - Rijndam Revalidatiecentrum, Rotterdam, South Holland

REFERENCES:
- [Derived] Dekker C, van Haastregt JCM, Verbunt JAMCF, de Jong JR, van Meulenbroek T, Pernot HFM, van Velzen AD, Bastiaenen CHG, Goossens MEJB. Pain-related fear in adolescents with chronic musculoskeletal pain: process evaluation of an interdisciplinary graded exposure program. BMC Health Serv Res. 2020 Mar 14;20(1):213. doi: 10.1186/s12913-020-5053-6. PMID 32171308
- [Derived] Dekker C, Goossens ME, Bastiaenen CH, Verbunt JA. Study protocol for a multicentre randomized controlled trial on effectiveness of an outpatient multimodal rehabilitation program for adolescents with chronic musculoskeletal pain (2B Active). BMC Musculoskelet Disord. 2016 Jul 28;17:317. doi: 10.1186/s12891-016-1178-5. PMID 27464953